CLINICAL TRIAL: NCT03410758
Title: Predictive Factors of Survival With and Without Repetition With 5 and 10 Years Curative Post-oesophagectomy for Cancer of the Oesophagus
Acronym: RESARPO
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: RESARPO
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2017-11

CONDITIONS: Esophageal Cancer; Esophageal Surgery Cancer; Overall Survival
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective study of Predictive Factors of Survival With and Without Repetition With 5 and 10 Years Curative Post-oesophagectomy for Cancer of the Oesophagus

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing during inclusion time carcinologic esophagectomy for esophageal cancer (Adenocarcinoma or epidermoid carcinoma)

Exclusion Criteria: Mortality within 90 postoperative days

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing esophagectomy for esophageal cancer
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France